CLINICAL TRIAL: NCT06770049
Title: Phenotype-Tailored Lifestyle Intervention for Obesity: A Randomized Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-002375; R01DK139028 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: In this 12-month, randomized, active-controlled trial, we aim to compare the effect of guiding lifestyle intervention tailored to a sub-classification of obesity based on physiological and behavioral alterations, called phenotypes.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Lifestyle Intervention (SLI) program (Active Comparator)
  Interventions: Behavioral: Standard Lifestyle Intervention (SLI) program
- Phenotype-tailored Lifestyle Intervention (PLI) program (Experimental)
  Interventions: Behavioral: Phenotype-tailored Lifestyle Intervention (PLI) program

INTERVENTIONS:
Behavioral: Standard Lifestyle Intervention (SLI) program — Subjects will receive recommendations for calorie and macronutrient intake, physical activity, and behavioral skills to be followed for 12 months and will be delivered by a multidisciplinary team of obesity experts in a 12-month structured follow up. Participants will meet with a registered dietician as well as member of the study team to learn more about their intervention. Diets will be prescribed for each participant with a 30% calorie deficit calculated from measured REE. Macronutrient composition will be guided based on the patient preference. Participants will be prescribed 150 minutes of physical activity per week (spread across 4-5 days) and recommendations to reach 10,000 steps daily. During the first 12 weeks, participants will be scheduled a 12-week behavioral program focusing on self-monitoring and stimulus control using cognitive-behavioral approaches to promote adherence to diet and exercise prescriptions.
  Arms: Standard Lifestyle Intervention (SLI) program
Behavioral: Phenotype-tailored Lifestyle Intervention (PLI) program — Subjects will receive recommendations for calorie and macronutrient intake, physical activity, and behavioral skills to be followed for 12 months and will be delivered by a multidisciplinary team of obesity experts. The recommendations will be determined a priori to tailor for each obesity phenotype
  Arms: Phenotype-tailored Lifestyle Intervention (PLI) program

SUMMARY:
The purpose of this study is to develop an evidence-based precision medicine approach for obesity that enhances weight loss and promotes weight loss maintenance.

ELIGIBILITY:
Inclusion:

• men or women between 18 to 65 years with obesity (BMI>30kg/m2).

Exclusion:

* weight change greater than 3% in the previous 3 months
* history of bariatric surgery and bariatric endoscopy
* untreated psychiatric disorders including binge eating disorders and bulimia
* current use of AOMs
* history of use of medications affecting weight or energy intake or energy expenditure in the last 6 months
* history of type 1 diabetes mellitus or uncontrolled medical conditions (e.g., uncontrolled hypertension)
* women who are pregnant or plan to become pregnant,
* any condition that limits their participation in the study
* Principal Investigator discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Total Body Weight Loss (TBWL) | Baseline, 52 weeks
  Change in Total Body Weight Loss (TBWL) in kg

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD,PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No